CLINICAL TRIAL: NCT00173381
Title: The Role of Lymphangiogenesis in Head and Neck Cancer Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700657
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-03-30 (Estimated); Status verified 2005-06

CONDITIONS: Oral Cancer; Laryngeal Cancer; Hypopharyngeal Cancer
Keywords: lymphangiogenesis; head and neck squamous cell carcinoma (HNSCC); vascular endothelial growth factor-C (VEGF-C); cyclooxygenase-2 (COX-2); interleukin-6 (IL-6)
MeSH Terms: conditions — Mouth Neoplasms; Laryngeal Neoplasms; Hypopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
The purpose of this study is to investigate the role of lymphangiogenesis in the metastasis of head and neck cancer.

DETAILED DESCRIPTION:
Head and neck cancer is a major, worldwide cause of morbidity and mortality. As long as the neoplasm is confined to its organ of origin, the patient can be cured through surgical removal of the tumor mass. Unfortunately, many cancers metastasize to other sites in the body, and metastasis is the leading cause of death in cancer patients. In principle, cancer cells can spread within the body by different mechanisms, such as direct invasion of surrounding tissues (per continuitatem), spread via the blood vascular system (hematogenous metastasis) and spread via the lymphatic system (lymphatic metastasis). Tumor cells can invade either the blood or lymphatic vessels to access the general circulation and then establish themselves in other tissues. Clinicopathological data suggest that the lymphatics are an initial route for the spread of solid tumors. Infiltration of lymphatic vessels by tumor cells has been found at the periphery of many experimental and human tumors, and the lymphatic system has been recognized as a conduit for tumor cell dissemination. Though the significance of angiogenesis for tumor progression has been well documented, the molecular mechanisms regulating the growth and function of lymphatic vessels are largely unknown.

Vascular endothelial growth factors, first identified in 1989, are well-known angiogenic agents and targets for anti-cancer therapies. Now it appears that VEGF-C, one recently-cloned member of the vascular endothelial growth factor (VEGF) family, is also involved in developmental and tumor-induced lymphangiogenesis. VEGF signals through two tyrosine kinase receptors, VEGFR-1 and VEGFR-2, which are expressed predominantly but not exclusively on vascular endothelial cells. As neither VEGFR-1 nor VEGFR-2 appears to be highly expressed in lymphatic endothelium, it was not surprising that a third VEGF receptor, VEGFR-3, was found to be predominantly expressed on lymphatic vessels during development. What was surprising, however, was that VEGF was not found to bind to VEGFR-3. Instead, VEGF-C was discovered to be ligand for VEGFR-3. Research groups provide direct evidence that VEGF-C is not only an important regulator of lymph vessel growth (lymphangiogenesis) in vivo but it also enhances lymphatic metastasis. Using experimental approaches, Mäkinen et al., Skobe et al., as well as Mandriota et al. demonstrate an important role of VEGFR-3 and its ligand, VEGF-C, in developmental and tumor-induced lymphangiogenesis. In normal adult human tissues, the VEGF-C receptor VEGFR-3 (FLT-4) is predominantly expressed by lymphatic endothelia. Expression of VEGF-C occurs in a variety of human tumors such as breast, colon, lung, thyroid, gastric, squamous cell cancers, mesotheliomas, neuroblastomas, sarcomas and melanomas. Moreover, expression of VEGF-C mRNA has recently been shown to correlate with the rate of metastasis to lymph nodes in breast, colorectal, gastric, thyroid, lung and prostate cancers. To date, however, lymphangiogenesis has not been causally linked to tumor metastasis.

Cyclooxygenase-2 (COX-2) enzyme catalyzes the synthesis of prostaglandins. COX-2 is an immediate-early response gene induced by inflammation, growth factors, tumor promoters, oncogenes, and carcinogens. Increased levels of COX-2 may contribute to carcinogenesis by modulating xenobiotic metabolism, apoptosis, immune surveillance, and angiogenesis. Any significant increase in tumor mass must be preceded by an increase in vascular supply to deliver nutrients and oxygen to the tumor. Recently, levels of COX-2 were found to correlate with both VEGF expression and tumor vascularization in HNSCC. This finding in human tissues is consistent with prior evidence that overexpression of COX-2 in epithelial cells led to enhanced production of VEGF and the formation of capillary-like networks. Although COX-2 contributes to the regulation of angiogenesis, its role in lymphangiogenesis is not clear.

IL-6 is a secreted, multifunctional glycoprotein. Through binding to α-chain (IL-6-R, gp80) and subsequently recruiting the β-chain (gp130) of the receptor, IL-6 performs various biological functions. The diversity of IL-6 signaling mediated via gp130 explains its functional pleiotropy. IL-6 regulates inflammatory reactions, immune responses, hepatic acute-phase protein synthesis, and several other important physiological processes. Interestingly, the influence of IL-6 in human cancers is varied depending on the cell types. For example, IL-6 has been demonstrated to promote growth of multiple myeloma, Kaposi's sarcoma, and prostatic cancer cells, while inhibiting the proliferation of lung and breast cancer cells. Previous investigations have confirmed that IL-6 is important in both physiological and pathological angiogenesis. Additionally, recent study supports the hypothesis that IL-6 facilitates tumorigenesis of cervical cancer via VEGF-mediated angiogenesis. Nevertheless, whether IL-6 could regulate the expression of VEGF-C and what is its role in lymphangiogenesis still need to be clarified.

Inhibition of angiogenesis is currently considered one of the most promising therapeutic strategies to inhibit cancer growth because it presumably can act on any tumor type, does not induce resistance of tumor cells (and can therefore be used in repeated therapeutic cycles) and has little effect on normal tissues. It now needs to be determined whether the same holds true for tumor lymphangiogenesis.

Metastases of head and neck cancers occur frequently through the lymphatic system, and the extent of lymph node involvement is a key prognostic factor for the diseases. In this study, we will conduct a systematic analysis of VEGF-C, COX-2 and IL-6 expressions and will try to find the correlation between their expressions, lymphatic metastases and patient survival. Next, we will investigate the relationship between VEGF-C, COX-2 and IL-6, and further clarify their effects on tumor growth. Undoubtedly, the findings of this study will help us understand whether lymphangiogenesis could be a focal point of anti-cancer research. If HNSCC tumors that express high levels of VEGF-C show a consistently higher incidence of lymphatic metastasis, then inhibition of VEGFR-3 function may be a novel approach to inhibit lymphatic metastasis in patients.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck squamous cell carcinoma

Exclusion Criteria:

* Other pathological type

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ting Tan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan